CLINICAL TRIAL: NCT03634124
Title: Generation of Thrombin and Prediction of Deep Vein Thrombosis Post Prosthetic Orthopedic Surgery of the Lower Limbs
Acronym: GT-PT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-01/ECN-01
Record Dates: First submitted 2018-08-07; First posted 2018-08-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2023-11

CONDITIONS: Deep Vein Thrombosis; Total Hip Prosthesis; Knee Prosthesis
MeSH Terms: conditions — Venous Thrombosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional group (Experimental)
  Interventions: Biological: Blood test; Other: Doppler ultrasound

INTERVENTIONS:
Biological: Blood test — Additional blood test of 4,5 ml of venous blood
Other: Doppler ultrasound — Vascular ultrasonic vascular exploration of the lower limbs

SUMMARY:
The numerical ratio between the value of the thrombin generation test performed without soluble thrombomodulin and the value of the thrombin generation test performed in the presence of soluble thrombomodulin, performed pre-surgically, could predict the risk of early venous thromboembolism after placement of total hip or knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have his consent and signed the consent form.
* The patient must affiliated or a beneficiary of a health insurance plan.
* The patient is at least 18 years old
* Patient with an indication of total hip prosthesis or total knee replacement surgery set unilateral

Exclusion Criteria:

* The patient is participating in another interventional study.
* The patient is in an exclusion period determined by a previous study.
* Minor patients, people in emergency situations.
* The patient is under the protection of justice, guardianship or curatorship.
* The patient refuses to sign the consent.
* It is not possible to inform the patient.
* The patient is pregnant, parturient, or breastfeeding.
* The patient has a contraindication (or incompatible drug combination) to drug thromboprophylaxis applied according to good clinical practice and recommendations of learned societies
* Long-term anticoagulant therapy for personal thrombotic history.
* Known hemorrhagic disease.
* Haemorrhagic risk perceived during the consultation of preoperative anesthesia, leading to modify / develop the usual thromboprophylaxis.
* Chronic liver disease.
* Chronic renal failure with calculated clearance <30 ml / min.
* Extreme body mass index: <18 kg.m-2 or> 40 kg.m-2
* total hip prosthesis or total knee prosthesis in the immediate aftermath of a bone fracture.
* total hip prosthesis resumption.
* Installation of more than one joint prosthesis.
* Surgery in the previous 3 months.
* Infective push in the previous 3 months.
* Indication of haemostatic treatment for abnormal haemorrhagic risk.
* Severe impairment of renal function with a calculated clearance <30 ml / min.
* Contraindication (allergic, metabolic, other ...) to usual drug thromboprophylaxis.
* Condition requiring dosage adjustment of drug thromboprophylaxis.
* Indication to put in place intermittent pneumatic compression for perioperative thromboprophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Estimate the numerical ratio between the value of the thrombin generation test performed without soluble thrombomodulin and the value of the thrombin generation test performed in the presence of soluble thrombomodulin | Day 0
  Numerical value
Occurrence of Symptomatic pulmonary embolism | Day 7 (± 2)
  yes/non
Occurrence of Symptomatic deep vein thrombosis somewhere in the body | Day 7 (± 2)
  Yes/no
Occurrence of Symptomatic deep vein thrombosis in legs | Day 7 (± 2)
  Yes/non

SECONDARY OUTCOMES:
Occurrence of proximal Symptomatic deep vein thrombosis in legs | Day 7 (± 2)
  Yes/no
Occurrence of distal Symptomatic deep vein thrombosis in legs | Day 7 (± 2)
  Yes/no
Occurrence of muscular Symptomatic deep vein thrombosis in legs | Day 7 (± 2)
  Yes/no
Occurrence of any kind of Symptomatic deep vein thrombosis in legs except muscular | Day 7 (± 2)
  Yes/no
Occurrence of proximal asymptomatic deep vein thrombosis in legs by doppler ultrasound | Day 7 (± 2)
  Yes/no
Occurrence of distal asymptomatic deep vein thrombosis in legs by doppler ultrasound | Day 7 (± 2)
  Yes/no
Occurrence of muscular asymptomatic deep vein thrombosis in legs by doppler ultrasound | Day 7 (± 2)
  Yes/no
Occurrence of any kind of asymptomatic deep vein thrombosis except muscular in legs by doppler ultrasound | Day 7 (± 2)
  Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Eva Cochery-Nouvellon, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Nimes University Hospital, Nîmes, France

REFERENCES:
- [Result] Chea M, Nouvellon E, Alonso S, Marchand P, Coulomb R, Kouyoumdjian P, Perin M, Laurent J, Mura T, Perez-Martin A, Bouvier S, Gris JC. Automated thrombin generation assay in patients entering hospital for total hip or knee arthroplasty: A prospective study. Thromb Res. 2026 Feb;258:109591. doi: 10.1016/j.thromres.2026.109591. Epub 2026 Jan 19. No abstract available. PMID 41570657